CLINICAL TRIAL: NCT06789536
Title: Evaluation of the Effectiveness of Routine Nurse Education in Prescribing Nicotine Replacement Therapy for Hospitalized Smokers in a University Hospital
Acronym: NICOTINURSE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: French National Cancer Institute (Institut National Du Cancer - France) (Unknown); Institut de Recherche en Santé Publique, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP241029
Record Dates: First submitted 2024-12-12; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Smoking Addiction
Keywords: Smoking; Addictology; Nicotine replacement therapy; Paramedical
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Intervention Model Description: Experimental Design:
  This is an open, cluster-randomized, stepped-wedge trial comparing smoking cessation rates at 1 month after hospital discharge between patients cared for by nurses trained in prescribing nicotine replacement therapies (NRTs) and those receiving standard care. In this design, departments are divided into 4 clusters, corresponding to nurse teams. At the start of the study, no team will have undergone training. Every 7 months, one team will be trained, with the training taking place over a 2-week period. Once a team is trained, the department will remain in the experimental group until the end of the study. No patients will be included in a department during its 2-week training period. The order in which departments undergo training will be randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trained nurses (Experimental): Nurses will participate in two one-hour training sessions, conducted in groups of three. This training will be provided by the smoking cessation team to learn how to prescribe nicotine replacement therapy, adjust dosages, and forward a referral letter to the patient's primary care physician and/or community nurse for continuity of care. They will receive a dosage adjustment guide to share with patients, along with the direct contact number for the smoking cessation team. Upon completing the training, nurses will be authorized to prescribe nicotine replacement therapy using the hospital's prescription software. Training will be spread over 15 days per department to avoid all nurses in the same unit being trained on the same day. Patients will receive information about nicotine replacement therapies and can try different formulations during hospitalization to optimize their choice. The outpatient addiction center team will be available to assist with any prescription-related questions.
  Interventions: Other: training nurses to prescribe nicotine substitutes, to adapt doses and to transmit to the outpatient physician and/or nurse nurse to facilitate the continuation of treatment
- No trained nurses (No Intervention): Physicians are informed about the intervention procedures of the Addiction Liaison Team (ELSA), accessible through a single central call number. Upon request, an ELSA team member visits the bedside of identified smoking patients, provides care recommendations to the attending physician, particularly regarding nicotine replacement therapy, and prescriptions are written by the patient's care team based on ELSA's guidance. ELSA maintains a standardized addiction care record to document recommendations, accessible to the healthcare team. During hospitalization, the team adjusts dosages, refers patients to addiction services or the Tobacco Info Service hotline upon discharge, and provides a nicotine replacement prescription with contact details for the patient's primary care providers. Discharge summaries written by patient's care team often include ELSA's recommendations to inform primary care physicians. Patients requesting continued care at HEGP are scheduled for follow-up appointment.

INTERVENTIONS:
Other: training nurses to prescribe nicotine substitutes, to adapt doses and to transmit to the outpatient physician and/or nurse nurse to facilitate the continuation of treatment — Nurses will undergo training sessions provided by the smoking cessation team to learn how to prescribe nicotine replacement therapy, adjust dosages, and forward a referral letter to the patient's primary care physician and/or community nurse for continuity of care. They will receive a dosage adjustment guide to share with patients. Upon completing the training, nurses will be authorized to prescribe nicotine replacement therapy using the hospital's prescription software.
  Arms: Trained nurses

SUMMARY:
The goal of this study is to determine whether training nurses to prescribe nicotine replacement therapy (NRT) can increase the proportion of smoking cessation at one month after hospital discharge among active smokers (daily or occasional tobacco use) hospitalized at the European Hospital Georges Pompidou in the following departments: Hypertension/Vascular Medicine, Nephrology, Pulmonology, and the Cardiac Intensive Care Unit.

The main questions it aims to answer are :

Does training nursing teams in the prescription and adjustment of nicotine replacement therapy increase the proportion of smoking cessation at one month after hospital discharge, defined as a total absence of tobacco consumption for at least seven days prior to the consultation, based on self-report and confirmed by an exhaled carbon monoxide (CO) level of ≤10 ppm? We will compare the usual care provided in the targeted departments with the care provided after all nurses in these departments receive training. The training will involve teaching the prescription of nicotine replacement therapy, dose adjustment, and communication with general practitioners and/or community nurses through a referral letter to facilitate continued care. Nurses will also have access to a dose adjustment document to provide to patients.

Participants will be followed up at discharge and at 1, 3, and 6 months post-discharge. At each visit, they will complete questionnaires on smoking behavior, quality of life, anxiety, and depression symptoms, and an exhaled CO measurement will be performed.

DETAILED DESCRIPTION:
Secondary questions it aims to answer are :

Does training nursing teams in the prescription and adjustment of nicotine replacement therapy :

* Reduce the average number of cigarettes smoked per day at 1, 3, and 6 months post-discharge?
* Decrease tobacco consumption by at least 50% at 1, 3, and 6 months post-discharge based on self-reported consumption?
* Increase the proportion of smoking cessation at 3 and 6 months post-discharge, defined as a total absence of tobacco consumption for at least seven days prior to the consultation, based on self-report and confirmed by an exhaled carbon monoxide level of ≤10 ppm?
* Improve patients' quality of life as measured by the SF-12 quality of life scale and symptoms of anxiety and depression assessed by the HAD scale at 1, 3, and 6 months post-discharge?
* Change the proportion of patients who access an addiction treatment center within six months post-discharge?
* Increase the use of nurse-prescribed nicotine replacement therapy during hospitalization and at discharge?
* Enhance nurse satisfaction with their practice?

ELIGIBILITY:
Inclusion Criteria:

* An active smoking patient (daily or occasional tobacco use) hospitalized in the following departments: hypertension/vascular medicine, nephrology, pulmonology, or the coronary care unit (CCU).
* Patient residing in the Île-de-France region.
* Proficient in the French language.
* Has signed informed consent.

Exclusion Criteria:

* Patient not affiliated with social security;
* Patient under State Medical Aid (AME);
* Patient under legal protection measures;
* Pregnant or breastfeeding patient;
* Patient refusing to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
smoking cessation one month after hospital discharge | 1 month after enrollment
  The primary outcome is smoking cessation one month after hospital discharge, defined as a total absence of tobacco use for at least 7 days prior to the consultation day, based on self-reported data and confirmed by an exhaled carbon monoxide measurement of 10 ppm or less.

SECONDARY OUTCOMES:
The average number of cigarettes smoked per day at 1, 3, and 6 months after hospital discharge | 1, 3 and 6 months after enrollment
  The average number of cigarettes smoked per day at 1, 3, and 6 months after hospital discharge based on self-reported data
The proportion of patients who reduced their consumption by at least 50% compared to their initial consumption | 1, 3, and 6 months after enrollment
  The proportion of patients who reduced their consumption by at least 50% compared to their initial consumption at 1, 3, and 6 months after hospital discharge, based on self-reported consumption.
The proportion of patients who achieved smoking cessation at 3 and 6 months after hospital discharge | 3 and 6 months after enrollment
  The proportion of patients who achieved smoking cessation at 3 and 6 months after hospital discharge, defined as a total absence of tobacco consumption for at least 7 days prior to the consultation day, based on self-reported data and confirmed by an exhaled carbon monoxide measurement of 10 ppm or less.
The patients' quality of life score | 1, 3, and 6 months after enrollment
  The patients' quality of life score measured using the 12-Item Short Form Survey (SF-12) quality of life scale available in the national smoking cessation consultation file published by Santé publique France, at 1, 3, and 6 months after hospital discharge. Minimum value of SF-12 is: 0, Maximum value is: 100 (representing the best possible health)
The patient's anxiety and depression | 1, 3, and 6 months after enrollment
  The patient's anxiety and depression measured using the Hospital Anxiety and Depression Scale (HAD) at 1, 3, and 6 months after hospital discharge. Minimum value is : 0, Maximum value: 42 (representing the worse possible)
The professional satisfaction score of nurses | Before the training and through study completion (41 months)
  The professional satisfaction score of nurses with a job satisfaction questionnaires that all nurses participating in the study will complete before the training and after the inclusion of the last patient. The minimum value is : 0 , maximal value : 40 (the best value)
Proportion of patients accessing an addiction center | 6 months after enrollment
  The proportion of patients who accessed an addiction center 6 months after hospital discharge.
The proportion of patients who received a nurse-prescribed nicotine replacement therapy (NRT) | During hospitalization (up to 2 months) and at discharge (up to 2 months)
  The proportion of patients who received a nurse-prescribed nicotine replacement therapy (NRT) during hospitalization and at discharge, measured through a data extraction from the prescription software, with the prescription being patient-specific and the nurse's authorization to prescribe recorded by the IT department.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Isabelle Tropeano, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (4):
- France (4):
  - Hôpital européen Georges-Pompidou - Hypertension artérielle et médecine vasculaire, Paris
  - Hôpital européen Georges-Pompidou - Néphrologie, Paris
  - Hôpital européen Georges-Pompidou - Pneumologie, Paris
  - Hôpital européen Georges-Pompidou - USIC, Paris

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered. The founder could be involved in the decision. Teams wishing obtain IPD must meet the sponsor and IP team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization. Processing of shared data must comply with European General Data Protection Regulation (GDPR).